CLINICAL TRIAL: NCT07044934
Title: Impact of Preoperative Uric Acid on Postoperative Acute Kidney Injury in Female Patients Undergoing Non-cardiac Surgery
Brief Title: Uric Acid and Menopausal Age in Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji-Hoon Sim, Assistant Professor, Asan Medical Center
Other Study IDs: AMC [2024-1090]
Record Dates: First submitted 2025-06-21; First posted 2025-07-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Uric Acid
Keywords: uric acid; female; non cardiac; acute kindeny injury; menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Premenopausal Women
  Interventions: Other: No Intervention: Observational Cohort
- Postmenopausal Women
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This observational cohort includes female patients undergoing non-cardiac surgery. No intervention was administered as part of the study protocol. Preoperative serum uric acid levels were measured, and patients were followed for the development of postoperative acute kidney injury. Data were analyzed retrospectively to assess the association between uric acid levels and acute kidney injury, with subgroup analyses based on menopausal status (premenopausal vs. postmenopausal women).

SUMMARY:
Preoperative serum uric acid significantly impacted acute kidney injury in female patients undergoing non-cardiac surgery, with differential effects observed before and after menopause.

DETAILED DESCRIPTION:
Preoperative serum uric acid has been increasingly recognized as a potential biomarker associated with acute kidney injury in various clinical settings. However, the sex-specific and hormonal influences on this association remain unclear, particularly in the context of non-cardiac surgery. Female patients, who experience significant physiological changes across the menopausal transition, may exhibit different renal susceptibilities to elevated serum uric acid levels.

In this retrospective cohort study, the investigators aimed to evaluate the association between preoperative serum uric acid levels and postoperative acute kidney injury in female patients undergoing non-cardiac surgery, with a particular focus on menopausal status. Women were stratified into premenopausal and postmenopausal groups based on age and clinical criteria. The investigators hypothesized that the threshold and pattern of serum uric acid-associated acute kidney injury risk may differ between these two populations due to differences in hormonal status and baseline renal reserve.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years and older who underwent elective non-cardiac surgery

Exclusion Criteria:

* Patients with gout
* Patients who underwent nephrectomy or kidney transplantation (either as recipients or donors)
* Patients diagnosed with chronic kidney disease or who had already undergone kidney replacement therapy
* Patients with estimated glomerular filtration rate < 30 mL/min/1.73m²; and patients with incomplete data or missing laboratory values

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This study included female patients aged 18 years or older who underwent elective non-cardiac surgery at a tertiary medical center. For patients who underwent multiple surgeries during the study period, only the first procedure following hospital admission was analyzed. The exclusion criteria were as follows: patients with a history of gout; those who had undergone nephrectomy or kidney transplantation (either as donors or recipients); patients diagnosed with chronic kidney disease or those who had received kidney replacement therapy; patients with an estimated glomerular filtration rate of less than 30 mL/min/1.73 m²; and those with incomplete clinical data or missing laboratory values.
Sampling Method: Non-Probability Sample
Enrollment: 127052 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Acute Kidney Injury | 7 days post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No
The dataset used and/or analyzed during the current study is available from the corresponding author upon reasonable request.